CLINICAL TRIAL: NCT04177095
Title: Immune Monitoring to Facilitate Belatacept Monotherapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Transplant Genomics, Inc. (Industry); CareDx (Industry)
Responsible Party: Principal Investigator, Hannah Gilligan, Principal investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019P002608
Record Dates: First submitted 2019-11-22; First posted 2019-11-26 (Actual); Results first posted 2023-12-04 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-12

CONDITIONS: Kidney Transplant Rejection; Immunosuppression
MeSH Terms: interventions — Abatacept; Mycophenolic Acid; Sirolimus; Everolimus; Prednisone

STUDY DESIGN:
Intervention Model Description: Prospective single-center, single-arm pilot study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Belatacept treated patients (Experimental): Renal transplant recipients treated with a combination of belatacept and any of the following: mycophenolate, sirolimus, everolimus and prednisone
  Interventions: Diagnostic Test: Allosure; Drug: Immunosuppression reduction; Diagnostic Test: Trugraf

INTERVENTIONS:
Diagnostic Test: Allosure — Monthly monitoring of dd-cfDNA levels in blood
  Other Names: donor-derived cell-free DNA (dd-cfDNA)
Drug: Immunosuppression reduction — Stepwise reduction in the dose, and ultimate discontinuation of, all non-belatacept immunosuppression (mycophenolate, sirolimus, everolimus, prednisone) guided by monitoring of Allosure and Trugraf results
  Other Names: Belatacept; mycophenolate; sirolimus; everolimus; prednisone
Diagnostic Test: Trugraf — Monthly monitoring of Trugraf result

SUMMARY:
* To determine the utility of novel blood-based immune monitoring tools (Allosure and Trugraf) to facilitate belatacept monotherapy.
* To determine the percent of belatacept-treated renal transplant patients that can be safely converted to belatacept monotherapy.

DETAILED DESCRIPTION:
This study will examine whether renal transplant recipients treated with a belatacept-based immunosuppressive regimen can safely be weaned off all non-belatacept immunosuppression (mycophenolate, mTORi, prednisone) in a stepwise fashion. To this end, participants will undergo monthly "immune monitoring" using the Allosure (dd-cfDNA) and Trugraf (RNA profiling) blood tests to determine if they are in a state of immune quiescence. Only patients who are deemed to be immune quiescent, will continue to be weaned of non-belatacept immunosuppression.

ELIGIBILITY:
Inclusion Criteria:

* Age minimum 18 years
* Written informed consent
* Single kidney transplant recipient (i.e. no combined organ transplants)
* Treated with de novo belatacept since transplantation (i.e. no previous use of calcineurin inhibitor or mTOR inhibitor for the current transplant)
* At least 1 year after transplantation or after initiation of belatacept
* Stable renal function (eGFR > 40 ml/min continuously during previous 6 months)
* Blood biomarkers indicate immune quiescence (for Allosure this corresponds to dd-cfDNA < 1%; for Trugraf this corresponds to "TX" signature)
* No history of BK viremia in current allograft

Exclusion Criteria:

* History of biopsy-proven acute rejection
* Presence of donor-specific antibodies (at any MFI)
* Spot urine protein/creatinine ratio > 0.5 g/g

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2023-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Gilligan, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Belatacept Treated Patients
Started | 17
Completed | 10
Not Completed | 7
Not completed — Withdrawal by Subject | 3
Not completed — Screen Failure | 3
Not completed — Problems with the Trugraf assay | 1

BASELINE CHARACTERISTICS:
Arm/Group | Belatacept Treated Patients
Number analyzed (Participants) | 17
Age, Customized [Count of Participants; unit: Participants]
  18 years or older | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 12
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Acute Rejection
Description: Biopsy-proven according to Banff 2017 criteria
Time Frame: Enrollment through 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Belatacept Treated Patients
Number analyzed (Participants) | 12
Participants | 0

2. Secondary Outcome: Increase in eGFR
Description: Calculated using CKD-EPI formula
Time Frame: From baseline to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Belatacept Treated Patients
Number analyzed (Participants) | 12
Participants | 6

3. Secondary Outcome: Rate of New-onset Proteinuria
Description: Defined as g/g creatinine, measured on random urine sample
Time Frame: At 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Belatacept Treated Patients
Number analyzed (Participants) | 12
Participants | 1

4. Secondary Outcome: Incidence of de Novo Donor Specific Antibodies
Description: Screened for using Luminex platform
Time Frame: At 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Belatacept Treated Patients
Number analyzed (Participants) | 12
Participants | 0

5. Secondary Outcome: Survival
Description: Overall and death-censored graft survival
Time Frame: At 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Belatacept Treated Patients
Number analyzed (Participants) | 12
Participants | 12

6. Primary Outcome: Incidence of Acute Rejection
Description: Biopsy-proven according to Banff 2017 criteria
Time Frame: Through study completion, 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Belatacept Treated Patients
Number analyzed (Participants) | 12
Participants | 0

ADVERSE EVENTS:
Time Frame: 2 Years
Arm/Group | Belatacept Treated Patients
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 5/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belatacept Treated Patients (N=12)
Urinary Tract Infection (Infections and infestations) | 1 (2)
Elevated LFTs (Investigations) | 1 (1)
Fatigue (Investigations) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Elevated Creatinine (Investigations) | 2 (2)
Knee Pain (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-25): https://cdn.clinicaltrials.gov/large-docs/95/NCT04177095/Prot_SAP_000.pdf